CLINICAL TRIAL: NCT05023187
Title: SCOT: An Online Intervention to Reduce Social Isolation and Promote Cognitive Well-being in the Elderly Population
Brief Title: Social and Cognitive Online Training: the SCOT Project
Acronym: SCOT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi di Trento (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Protocol 2020-036
Record Dates: First submitted 2021-06-14; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-04

CONDITIONS: Aging; Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social and Cognitive Online Training Group (SCOT) (Experimental): A group of participants randomly assigned to a social-cognitive online training through individual cognitive training sessions and group sessions to improve social functioning.
  Interventions: Behavioral: SCOT
- Control Group (CON) (Active Comparator): A group of participants randomly assigned to receive an active control intervention to compare performances with the experimental group.
  Interventions: Behavioral: CON

INTERVENTIONS:
Behavioral: SCOT — A 8-week social and cognitive online training to improve both cognitive and social functioning, which includes 2 sessions (~45 minutes each) of individual cognitive training through the BrainHQ© program 2020 (BrainHQ© Posit Science) and a psycho-educational group session for each week (24 sessions in total).
  In the experimental intervention, all activities are focused on enhancing executive functions (working memory, processing speed, inhibitory control etc.) and social cognition abilities (identifying/recognizing facial expressions, styles attribution, drawing conclusions etc.).
  Arms: Social and Cognitive Online Training Group (SCOT)
Behavioral: CON — A 8-week active control intervention consisting of 2 sessions (~45 minutes each) of cognitive stimulation exercises and a group session for each week (24 sessions in total) during which the various cognitive domains are deepened and the exercises carried out during the week are reviewed all together.
  The online control intervention has been specifically designed to increase the cognitive involvement of the subjects and to replicate the condition of exposure to social dynamics.
  Arms: Control Group (CON)

SUMMARY:
Social isolation and reduced involvement in cognitive activities are associated with repercussions on cognitive well-being and health status in elderly adults. In particular, loneliness and social isolation represent risk factors in favouring cognitive decline and dementia. The Social Cognition Online Training (SCOT) project aims to evaluate the beneficial effects of an online intervention on social-cognitive functioning in healthy elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* Cognitively healthy subjects aged above 65 years old
* Montreal Cognitive Assessment (MoCA) equivalent score > 1 (Italian normative values)

Exclusion Criteria:

* Diagnosis of dementia, based on Diagnostic and Statistical Manual of Mental Disorders, FifthEdition (DSM-V)
* History of current or previous neuropsychiatric disorders;
* History of current or previous substance abuse;

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-19 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
The Tower of London test (Boccia et al. 2017) | Day 0 - Month 3
  Accuracy (% of correct answers)

SECONDARY OUTCOMES:
Experimental task of emotion recognition | Day 0 - Month 3
  Accuracy (% of correct answers)
Italian Social and Emotional Loneliness Scale | Day 0 - Month 3
  Minimum value: 18; Maximum value: 72; Higher scores mean a worse outcome in terms of perceived loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: Costanza Papagno, Study Director — Centro Interdipartimentale Mente/Cervello - CIMeC; Alessandra Dodich, Principal Investigator — Centro Interdipartimentale Mente/Cervello - CIMeC
Locations (1):
- Centro Interdipartimentale Mente/Cervello - CIMeC, Rovereto, Trento, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Funghi G, Meli C, Cavagna A, Bisoffi L, Zappini F, Papagno C, Dodich A. The Social and Cognitive Online Training (SCOT) project: A digital randomized controlled trial to promote socio-cognitive well-being in older adults. Arch Gerontol Geriatr. 2024 Jul;122:105405. doi: 10.1016/j.archger.2024.105405. Epub 2024 Mar 5. PMID 38531149